CLINICAL TRIAL: NCT06837272
Title: A Longitudinal Study to Explore the Impact of Gut Microbiome on Brain Health in Alzheimer's Disease: China Healthy Brain and Gut Microbiome Study (CHBGMS)
Brief Title: A Longitudinal Study to Explore the Impact of Gut Microbiome on Brain Health in Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Jining Medical University (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Can Sheng, Professor, Jining Medical University
Other Study IDs: JiningMU_Shc1
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Gut Microbiota; Metabonomics; Magnetic Resonance Imaging
Keywords: Subjective cognitive decline; Multi-omics
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — In this project, the investigators will test ApoE genotype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cognitively normal group: (1) normal performance on standardized cognitive tests; (2) with no cognitive complaints or any concerns (worries).
- Subjective cognitive decline (SCD) group: (1) self-experienced persistent decline in memory, rather than other domains of cognition; (2) normal performance on standardized cognitive tests; (3) failure to meet the criteria for MCI or dementia; (4) age at onset of SCD ≥ 60 years old; (5) onset of SCD within the last 5 years; (6) concerns (worries) associated with SCD; (7) feeling of worse performance than others of the same age group.
  Interventions: Diagnostic Test: Multi-omics features extraction
- Mild cognitive impairment (MCI) group: (1) having impaired scores on both measures in at least one cognitive domain (memory, language, or speed/executive function); (2) having impaired scores in each of the three cognitive domains (memory, language, or speed/executive function); (3) the Functional Activities Questionnaire (FAQ)≥9.
- AD dementia group: (1) meet the criteria for dementia and have impaired daily functional activities; (2) episodic memory deficit; 3) Clinical Dementia Rating (CDR) ≥ 1.

INTERVENTIONS:
Diagnostic Test: Multi-omics features extraction — Based on multi-omics features extracted from clinical data, gut microbiome, metabolomics, and multi-modal MRI, the diagnostic model of SCD due to preclinical AD will be established.
  Groups: Subjective cognitive decline (SCD) group

SUMMARY:
Gut microbiota dysfunction is associated with Alzheimer's disease (AD). However, the potential modulatory mechanism remains unclear. Previous studies have shown that gut-derived metabolites short-chain fatty acids (SCFAs) may be the key mediators between gut microbiota and brain, participating in the modulatory pathway "gut microbiota-SCFAs-brain networks". In this project, high-throughput targeted metabolomics technique will be used to explore the differences of SCFAs in the spectrum of AD, including cognitively normal individuals, subjective cognitive decline (SCD), mild cognitive impairment (MCI), and AD dementia. Then, the gut microbiome and multi-modal MRI techniques will be combined to elucidate potential interaction mechanisms of "gut microbiota-SCFAs-brain networks". Finally, based on multi-omics features extracted from gut microbiome, metabolomics, and neuroimaging after five years, the diagnostic model of SCD due to preclinical AD will be established using machine learning methods.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively normal group:

  1. normal performance on standardized cognitive tests;
  2. with no cognitive complaints or any concerns (worries).
* SCD group:

  1. self-experienced persistent decline in memory, rather than other domains of cognition;
  2. normal performance on standardized cognitive tests;
  3. failure to meet the criteria for MCI or dementia;
  4. age at onset of SCD ≥ 60 years old;
  5. onset of SCD within the last 5 years;
  6. concerns (worries) associated with SCD;
  7. feeling of worse performance than others of the same age group.
* MCI group:

  1. having impaired scores on both measures in at least one cognitive domain (memory, language, or speed/executive function);
  2. having impaired scores in each of the three cognitive domains (memory, language, or speed/executive function);
  3. the Functional Activities Questionnaire (FAQ)≥9.
* AD dementia group:

  1. meet the criteria for dementia and have impaired daily functional activities;
  2. episodic memory deficit; 3) Clinical Dementia Rating (CDR) ≥ 1.

Exclusion Criteria:

* a history of stroke;
* major depression and anxiety;
* other central nervous system disorders that may cause cognitive impairment, such as Parkinson's disease, tumors, encephalitis, and epilepsy;
* cognitive impairment caused by traumatic brain injury;
* systemic diseases, such as thyroid dysfunction, syphilis and HIV;
* psychosis or congenital mental developmental delay;
* a history of using antibiotics, probiotics, prebiotics, or synbiotics within 3 months;
* the use of corticosteroid, immune stimulating medications, and immunosuppressive agents;
* major gastrointestinal tract surgery in past 5 years;
* severe gastrointestinal diseases, such as irritable bowel syndrome, infammatory bowel disease, severe gastritis, other dysfunction in digestion and absorption, which has been reported to infuence gut microbiota

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers recruited from both clinical and communities, and signed up with informed consent.
Sampling Method: Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes of gut microbiome in the spectrum of AD | 5 year
  Using the 16S rRNA Illumina Miseq sequencing technique, the diversity and compositions of gut microbiome will be compared in different stages of AD, including cognitively normal individuals, SCD, MCI and AD dementia.
The changes of SCFAs in the spectrum of AD | 5 year
  Using the high-throughput target metabolomics technique, SCFAs will be compared in different stages of AD, including cognitively normal individuals, SCD, MCI and AD dementia.
Multi-omics biomarkers associated with conversion to cognitive impairment for SCD subjects | 5 years
  SCD subjects will be followed for five years. The investigators aim to characterize those who convert to MCI or AD dementia during the follow-up, and further find the multi-omics features associated with the progression of AD. Based on multi-omics features extracted from clinical data, gut microbiome, metabolomics, and multi-modal MRI, the diagnostic model of SCD due to preclinical AD will be established.

SECONDARY OUTCOMES:
The interaction mechanisms of "gut microbiota-SCFAs-brain networks" | 5 years
  The gut microbiome, SCFAs and multi-modal MRI techniques will be combined to elucidate potential interaction mechanisms of "gut microbiota-SCFAs-brain networks".

CONTACTS AND LOCATIONS:
Overall Officials: Can Sheng, PhD, Principal Investigator — Jining Medical University
Locations (1):
- Department of Neurolgy, the Affiliated Hospital of Jining Medical University, Jining, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
The information of neuropsychological tests, and other clinical data are to be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: When summary data are published or starting 12 months after publication.
Access Criteria: When summary data are published or starting 12 months after publication.